CLINICAL TRIAL: NCT05101148
Title: A Phase I, Single-Arm, Sequential Study to Evaluate the Effect of Food on the Gastrointestinal Tolerability and Pharmacokinetics of Selumetinib After Multiple Doses in Adolescent Children With Neurofibromatosis Type 1 Related Plexiform Neurofibromas
Brief Title: Phase I Study to Assess the Effect of Food on the PK and Gastrointestinal Tolerability of Selumetinib in Adolescent Children With Neurofibromatosis Type 1 Related Plexiform Neurofibromas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1346C00015; 2024-517216-29-00 (Registry Identifier: EU (CTIS)); 2020-005648-52 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-11-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- selumetinib single arm (Experimental): This is a sequential study consisting of a screening period lasting up to 28 days, a 28 day (1 cycle) treatment period (T1) in a fed state, a 7 day washout period, a further 1 cycle treatment period (T2) in a fasted state and an extension to T2 until results from the primary analysis are available. During Treatment Period 1 and 2 all participants will receive selumetinib (25 mg/m2 bid). If a third treatment period (T3) is required, participants will enter a 7 day washout period followed by a treatment period in a fed state at an adjusted dose for 3 cycles.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — The dosing regimen for selumetinib (25 mg/m2 bid) will be based on BSA, during T1 and T2 the dose will be 25mg/m2, consistent with the approved prescribing information in the US. If T3 is required, appropriate dose of selumetinib will be defined by Data Review Committee for T3.

SUMMARY:
This study in adolescent participants with NF1 who have inoperable PN is designed to evaluate the effect of a low fat meal on steady state selumetinib exposure; to assess the effect on GI tolerability when selumetinib is dosed under fed and fasted conditions; and potentially, to confirm an appropriate dosing recommendation of selumetinib with a low fat meal that maintains efficacy with acceptable safety. These results may support labelling statements with regard to posology and food.

DETAILED DESCRIPTION:
Selumetinib is approved by the FDA for the treatment of paediatric patients 2 years of age and older with NF1 who have symptomatic, inoperable PN.

The efficacy of selumetinib in the treatment of NF1 related inoperable PN in paediatric participants was demonstrated in the SPRINT study in which selumetinib was taken at 25 mg/m2 bid under fasted conditions (fast for 2 hours before each dose and 1 hour after each dose). Safety data from this study showed that selumetinib has a generally predictable and manageable safety profile in this population. Gastrointestinal AEs were commonly reported but were predominantly mild/moderate in severity, predictable, and generally did not affect the ability of participants to remain on treatment. However, GI AEs in this paediatric study were reported at a higher frequency than that reported in an analysis of selumetinib in adult oncology participants. Dosing in a fed state is known to reduce GI tolerability for some oncology drugs; such a dosing regimen has an added benefit of improving compliance and adherence to dosing posology.

Food-effect studies conducted in healthy participants (Study D1532C00069) and adult participants with cancer (Study D1532C00020) show that consumption of a high fat meal reduces absorption of selumetinib: in healthy participants Cmax was reduced by 50% and AUC by 16%; and in participants with cancer Cmax was reduced by 62% and AUC by 19%. A further study in adult healthy participants (D1532C00089) found that a low fat, low calorie meal reduces the rate of absorption (Cmax reduced by 65% and tmax delayed by 2.5 hours) and the extent of absorption (AUC reduced by 38%) after a single dose of selumetinib. The finding that a low fat meal had a greater impact on exposure than a high fat meal is unusual and without a clear explanation although in vitro dissolution data suggest that the capsule shell disintegration may be impacted by food.

The study is designed to evaluate the steady state systemic exposure and safety (especially GI tolerability) of selumetinib 25 mg/m2 bid given with a low fat meal versus the same dose given in a fasted state. A third treatment period (T3) will be initiated if there is a significant reduction in exposure (AUC0-12, SS between T2 vs T1) when selumetinib is given with a low fat meal compared with a fasted state; T3 will evaluate the PK and safety of an adjusted dose of selumetinib when given with a low fat meal. The recommendation as to whether to initiate T3, and the dose to be used in T3, will be made by a DRC. This recommendation will be reviewed with FDA before dosing in T3 is initiated.

Approximately 20 participants will be enrolled to achieve 16 evaluable participants completing T2. An evaluable participant is defined as having received study treatment and provided the last required PK sample in T2.

A Data Review Committee(DRC) will review the PK and safety data from T1 and T2 and determine whether T3 is required. If T3 is required the DRC will select the dose to be used. The recommendation will be reviewed with FDA before dosing in T3 is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥ 12 to < 18 years at the time of signing the informed consent.
* All study participants must be diagnosed with (i) NF1 per NIH Consensus Development Conference Statement and (ii) inoperable PN. In addition to PN, participants must have at least 1 other diagnostic criterion for NF1 as defined in protocol.
* Participants must require treatment for NF1 and inoperable PN due to actual symptoms or because of the potential to develop significant clinical complications, as judged by the Investigator, as defined in the protocol.
* Participants who have had prior treatment with any MEKi (including selumetinib) may be considered for inclusion in this study.
* Participants must have a BSA ≥ 1.3 and ≤ 2.5 m2

Exclusion Criteria:

* Evidence or suspicion of optic glioma, malignant glioma, MPNST, or other cancer requiring treatment with chemotherapy or radiation therapy
* Prior malignancy requiring active treatment (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the participant had been disease free for ≥ 2 years or which would not have limited survival to < 2 years).
* A life-threatening illness, medical condition, organ system dysfunction of laboratory finding which, in the Investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of selumetinib, or put the study outcomes at undue risk.
* Participants with clinically significant cardiovascular disease as listed in the protocol.
* Liver function tests: bilirubin > 1.5 × the ULN for age (with the exception of those with Gilbert syndrome) or AST/ALT > 2 × upper limit of normal.
* Renal Function: Creatinine clearance or radioisotope glomerular filtration rate < 30 mL/min/1.73 m2 or a serum creatinine > 1.2 mg/dL (for participants aged between 12 and 15 years) or > 1.5 mg/dL for participants aged > 15 years).
* Participants with abnormal ophthalmological findings/conditions as listed in the protocol.
* Have any unresolved chronic toxicity, associated with previous therapy for NF1-PN: Gastrointestinal toxicity of CTCAE Grade 1 or higher; Have any other unresolved chronic toxicity with CTCAE Grade ≥ 2, except hair changes (such as alopecia or hair lightening).
* Participants who have previously been treated with a MEKi (including selumetinib) and either discontinued treatment or required a dose reduction due to toxicity
* Have had recent major surgery within a minimum of 4 weeks prior to starting study intervention, with the exception of surgical placement for vascular access. Have planned major surgery during the treatment period.
* Any multivitamin containing vitamin E must be stopped at least 7 days prior to initiation of selumetinib.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Selumetinib area under the plasma concentration-time curve from zero to 12 hours post-dose (AUC0-12) | At pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose (Cycle 1 Day 8 of each treatment period 1, 2 and 3); Each treatment period 1 and 2 has 1 cycle (Each cycle is 28 days). If needed, treatment period 3 will be started approximately 5 cycles later.
  To compare the AUC0-12, SS of the fed (same dose and dose adjustment if necessary) versus fasted state
Gastrointestinal Adverse Events graded by CTCAE Ver 5.0 (Grade 1 to 5) | from screening until 30 days after last dose
  To investigate the gastrointestinal toxicities of selumetinib capsules after multiple doses
Assessing change of Gastrointestinal toxicity diary: Modified Bristol Stool Form Scale for Children (mBSFS-C) | At screening (at least 14 days), Cycle 1 of each treatment period 1, 2 and 3 (1 cycle is 28 days)
  To investigate the gastrointestinal toxicities of selumetinib capsules after multiple doses
Assessing change of Gastrointestinal toxicity diary: Nausea and Vomiting Symptom Rating Scale (adapted from the Children's Cancer and Leukaemia Group) | At screening (at least 14 days), Cycle 1 of each treatment period 1, 2 and 3 (1 cycle is 28 days)
  To investigate the gastrointestinal toxicities of selumetinib capsules after multiple doses
Number of patients who take each gastrointestinal medication | From screening until 30 days after last dose
  Collecting gastrointestinal concomitant medications taken including, but not restricted to, medications used to treat diarrhoea, nausea and vomiting.
Proportion of patients who take each gastrointestinal medication | From screening until 30 days after last dose
  Collecting gastrointestinal concomitant medications taken including, but not restricted to, medications used to treat diarrhoea, nausea and vomiting.

SECONDARY OUTCOMES:
Adverse events(AEs) graded by CTCAE Version 5.0 | From screening until 30 days after last dose
  To further assess the safety and tolerability of selumetinib capsules
Maximum Peak plasma concentration (Cmax) of selumetinib and N-desmethyl selumetinib | At pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose (Cycle 1 Day 8 of each treatment period 1, 2 and 3); Each treatment period 1 and 2 has 1 cycle (Each cycle is 28 days). If needed, treatment period 3 will be started approximately 5 cycles later.
  To further evaluate the PK of selumetinib and N-desmethyl selumetinib metabolite after multiple doses under fed conditions, compared to fasted conditions
Area under the concentration-time curve from time zero to time of last measurable concentration (AUClast) of selumetinib and N-desmethyl selumetinib | At pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose (Cycle 1 Day 8 of each treatment period 1, 2 and 3); Each treatment period 1 and 2 has 1 cycle (Each cycle is 28 days). If needed, treatment period 3 will be started approximately 5 cycles later.
  To further evaluate the PK of selumetinib and N-desmethyl selumetinib metabolite after multiple doses under fed conditions, compared to fasted conditions
Time to maximum concentration (tmax) of selumetinib and N-desmethyl selumetinib | At pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose (Cycle 1 Day 8 of each treatment period 1, 2 and 3); Each treatment period 1 and 2 has 1 cycle (Each cycle is 28 days). If needed, treatment period 3 will be started approximately 5 cycles later.
  To further evaluate the PK of selumetinib and N-desmethyl selumetinib metabolite after multiple doses under fed conditions, compared to fasted conditions
Time to last measurable concentration (tlast) of selumetinib and N-desmethyl selumetinib | At pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose (Cycle 1 Day 8 of each treatment period 1, 2 and 3); Each treatment period 1 and 2 has 1 cycle (Each cycle is 28 days). If needed, treatment period 3 will be started approximately 5 cycles later.
  To further evaluate the PK of selumetinib and N-desmethyl selumetinib metabolite after multiple doses under fed conditions, compared to fasted conditions

CONTACTS AND LOCATIONS:
Overall Officials: Study physician Study physician, MD, Study Director — AstraZeneca
Locations (8):
- United States (2):
  - Research Site, Rochester, Minnesota
  - Research Site, Akron, Ohio
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Warsaw
- Research Site, Moscow, Russia
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Viskochil D, Wysocki M, Learoyd M, Sun P, So K, Evans A, Lai F, Hernandez HS. Effect of food on selumetinib pharmacokinetics and gastrointestinal tolerability in adolescents with neurofibromatosis type 1-related plexiform neurofibromas. Neurooncol Adv. 2024 Mar 16;6(1):vdae036. doi: 10.1093/noajnl/vdae036. eCollection 2024 Jan-Dec. PMID 38721358
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1346C00015&attachmentIdentifier=d1f9337d-eb8f-4b6d-9219-9d5724c9064a&fileName=D1346C00015_Synopsis_Redacted.pdf&versionIdentifier=